CLINICAL TRIAL: NCT07109674
Title: Inelastic Compression With a High Stiffness Index in Breast Cancer-related Lymphedema: A Prospective Case - Control Study
Brief Title: Adjustable Compression Wraps (ACW) in Lymphedema
Acronym: ACW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 345/BS/IRK/2024
Record Dates: First submitted 2025-06-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema; Lymphedema Arm; Breast Cancer
Keywords: breast cancer survivors; compression therapy; adjustable compression wrap; compression bandaging
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison the physiotherapeutical intervention in breast cancer surivors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjustable compression wrap-reduction kit (Experimental): The objective of this study was to compare the effectiveness on volume reduction, physical functioning and comfort of inelastic compression: adjustable compression wrap (reduction) at the intensive phase of treatment in advanced upper limb lymphedema among breast cancer survivors
  Interventions: Device: adjustable compression device (type circaid® reduction kit, Medi-Bayreuth)
- Compression bandaging (Active Comparator): text
  Interventions: Device: Comparison of inelastic compression efficiency

INTERVENTIONS:
Device: adjustable compression device (type circaid® reduction kit, Medi-Bayreuth) — inelastic compression during intensive phase of physical therapy
  Other Names: compression therapy
  Arms: Adjustable compression wrap-reduction kit
Device: Comparison of inelastic compression efficiency — The effect of compression on volume reduction, physical functioning, disease-related symptoms and comfort
  Arms: Compression bandaging

SUMMARY:
Compression therapy based on multilayer compression bandaging and com pression garment use remains the most efficient component of complex physical therapy (CPT) in lymphedema treatment. The proper self-application of compression bandages is generally considered as problematic. Adjustable compression wraps (ACW) have been proposed as an alternative to the commonly used short-stretch bandages for lymphedema. These systems allow easy application and removal for patients. They have been tested in patients with vascular disorders of the lower limbs and can be considered in breast cancer survivors with upper-limb lymphedema.

The objective of this study was to compare the effectiveness, physical functioning and comfort of 2 types inelastic compression: adjustable compression wrap (reduction) and multi-layer compression bandaging at the intensive phase of treatment in advanced upper limb lymphedema among breast cancer survivors.

DETAILED DESCRIPTION:
55 women after breast cancer treatment admitted to the Lymphedema Clinic and patients fulfilled the admission criteria - stage-II (according to ISL) lymphedema, ≥20% excess limb volumes, positive pitting skin sign, and absent signs of active cancer, venous thrombosis or previous compression were assigned into the experimental group with the adjustable compression wrap redcution kit, ACW - Group or the control with compression bandaging, CB-Group.

In the ACW reduction group, adjustable compression garments (typ circaid® reduction kit, Medi-Bayreuth) was also fitted based on individual limb measurements with ability to reduce size of garment as the limb volume decreases. The kit included a card with a color scale that allowed users to achieve the appropriate pressure of 20-30 mmHg. The next day, in order to refresh and moisturize the skin, these products were removed for a short period prior to the next therapeutic session. They were used for 24 hours.

In the CB group, multi-layer bandaging of the limb was performed using short stretch bandages with pads (Rosidal K, Lohmann & Raucher). At the beginning of bandaging, a cotton tube stockinet was placed on the arm, a layer of gauze was applied to the fingers and hand. A layer of foam padding (Lymphset: Lohmann & Raucher) was placed on the hand and wrapped around the arm. Three bandages of different sizes (8, 10, 12 cm in width) were placed around the limb with the first starting at the hand, the second at the wrist and the third beginning below the elbow. Sub-bandage pressure was measured via the Kikushime device (Kikgel, Ujazd Poland) on the dorsal part of the forearm, as well as on the arm, to ensure a pressure value within the range of 20-30 mmHg, comparable to pressure used in the compression system among the ACW Group. Bandages were removed for a short time before the therapeutic session the next day, as in the ACW-Group, and put on the next day. The exercise program including aerobic exercises of the upper limbs combined with deep breathing was performed in adjustable compression wraps or bandaging for 15 minutes in 1 session per day.

Measurements, including physical functioning, limb volumes and disease-related symptoms, were performed before the intervention and after treatment in both groups. Circumferential upper limb measurements were taken with the arm abducted at 30°, starting at the level of the ulnar styloid, every 4 cm proximal to this point along both limbs. Calculation of limb segment volumes was carried out using a simplified frustum formula (summed truncated cone). The excess volume was the difference between the affected and unaffected limbs expressed in litres. The percentage reduction of the excess volume was obtained as follows: (excess volume before treatment - excess volume after treatment) x 100/excess volume before treatment.

Patients rated their physical functioning, disease-related symptoms, compression comfort and complications of compression on a numerical rating scale (NRS) based on the International Compression Club (ICC) Questionnaire - Part for Patients. Firstly, the patients assessed their physical functioning (sum of ability to move wrist, elbow, shoulder; use a spoon; carry out work; complete household chores; practice sports' carry out leisure activities; social activities, on the Number Rating Scale (NRS; 0 = not able at all, 10 = completely able) and disease-related symptoms (sum of pain; loss of muscle strength; heaviness; swelling; tight skin; tingling; leakage; NRS: 0 = no complaints, 10 = the highest intensity), first without the tested compression and continued after 1 and 2 weeks using the compression device. Complications of compression related to skin irritation; tender spots; skin damage; itching; warmth; throbbing; cramps; cutting in; slippage; local swelling; bulky feeling; too tight feeling (NRS: 0 = not present at all, 10 = very obviously present, sum of points) were assessed after 1 and 2 weeks in both groups. Compression comfort including: easy donning; easy doffing; feeling immediately after donning; feeling during daytime; putting on clothes on compression; feeling at night; the appearance of the garment (NRS: 0 = not able at all, 10 = completely able, sum of points) was evaluated after the first and second weeks in both groups.

Treatment in both groups lasted 10 days (2 weeks, Monday to Friday). In the first week, all patients were treated by 2 experienced physiotherapists and educated in applying adjustable compression wraps (ACW reduction group) or self-bandaging (CB group). During the 2nd week, the use of ACW and CB was continued by the patients themselves at home. Patients were asked to maintain the adjustable compression wraps or compression bandaging even during the weekend (Saturday and Sunday).

ELIGIBILITY:
Inclusion Criteria:

* stage-II of lymphedema (according to ISL)
* ≥20% excess limb volumes
* positive pitting skin sign
* absent signs of active cancer
* absent of venous thrombosis

Exclusion Criteria:

* active cancer during oncological treatment
* using compression
* stage-I of lymphedema (according to ISL)
* < 20 % excess limb volumes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
The assessment of limb volume | 14 months
  Measurements including limb volumes were performed before the intervention, and after treatment in both groups. Circumferential upper limb measurements were taken with the arm abducted at 30°, starting at the level of the ulnar styloid, every 4 cm proximal to this point along both limbs. Calculation of limb segment volumes was carried out using a simplified frustum formula (summed truncated cone). The excess volume was the difference between the affected and unaffected limbs expressed in litres. The percentage reduction of the excess volume was obtained as follows: (excess volume before treatment - excess volume after treatment) x 100/excess volume before treatment.
The assessment of physical functioning | 14 months
  Patients rated their physical functioning of the affected limb on a numerical rating scale (NRS) based on the International Compression Club (ICC) Questionnaire - Part for Patients. The patients assessed their physical functioning (sum of ability to move wrist, elbow, shoulder; use a spoon; carry out work; complete household chores; practice sports' carry out leisure activities; social activities, on the Number Rating Scale (NRS; 0 = not able at all, 10 = completely able) before and after treatment in both groups.
The assessment of disease - related symptoms | 14 months
  Patients rated their disease-related symptoms based on the International Compression Club (ICC) Questionnaire - Part for Patients on the Number Rating (sum of pain; loss of muscle strength; heaviness; swelling; tight skin; tingling; leakage; NRS: 0 = no complaints, 10 = the highest intensity) before the intervention and after treatment in both groups.
The assessment of compression comfort | 14 months
  Patients rated their comfort and complications related to compression on a numerical rating scale (NRS) based on the International Compression Club (ICC) Questionnaire - Part for Patients. Complications of compression related to skin irritation; tender spots; skin damage; itching; warmth; throbbing; cramps; cutting in; slippage; local swelling; bulky feeling; too tight feeling (NRS: 0 = not present at all, 10 = very obviously present, sum of points) were assessed after treatment in both groups. Compression comfort including: easy donning; easy doffing; feeling immediately after donning; feeling during daytime; putting on clothes on compression; feeling at night; the appearance of the garment (NRS: 0 = not able at all, 10 = completely able, sum of points) was evaluated after treatment in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University School of Physical Education, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: Yes
* limb volume reduction
  * physical functioning
  * disease- related symptoms
  * comfort in compression
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after publication start date: 01.10.2025 end date: 31.12.2025
Access Criteria: IPD will be available to reviewers of the manuscript submitted for publication.
URL: https://www.akf.krakow.pl/

REFERENCES:
- [Background] Ochalek K, Kurpiewska J, Gradalski T. Adjustable Compression Wraps (ACW) vs. Compression Bandaging (CB) in the Acute Phase of Breast Cancer-Related Arm Lymphedema Management-A Prospective Randomized Study. Biology (Basel). 2023 Mar 31;12(4):534. doi: 10.3390/biology12040534. PMID 37106735
- [Background] Pujol-Blaya V, Salinas-Huertas S, Catasus ML, Pascual T, Belmonte R. Effectiveness of a precast adjustable compression system compared to multilayered compression bandages in the treatment of breast cancer-related lymphoedema: a randomized, single-blind clinical trial. Clin Rehabil. 2019 Apr;33(4):631-641. doi: 10.1177/0269215518821785. Epub 2019 Jan 4. PMID 30607986
- See also: Effectiveness of a precast adjustable compression system compared to multilayerd compression bandaging in the treatment of breast cancer-related lymphedema — https://pubmed.ncbi.nlm.nih.gov/37106735/